CLINICAL TRIAL: NCT01422499
Title: Phase I/II Intra-patient Dose Escalation Study of Vorinostat in Children With Relapsed Solid Tumor, Lymphoma or Leukemia
Brief Title: Vorinostat in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: University Hospital Heidelberg (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2007-11-02-1004
Record Dates: First submitted 2011-08-03; First posted 2011-08-24 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Children With Relapsed Solid Tumor, Lymphoma or Leukemia
Keywords: pediatric oncology; relapsed solid tumor; lymphoma; leukemia; vorinostat
MeSH Terms: conditions — Lymphoma; Leukemia | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: zolinza/vorinostat — orally once per day (suspension of 50mg/ml or capsules of 100 mg vorinostat); starting dose will be 180 mg/m²/d; escalated with increments of 50 mg/m²/d every two weeks until dose limiting toxicity (grade 3 or 4 toxicity according to CTC) occurs or up to a maximum dose of 580 mg/m²/d; This dose will then be applied for 3 months. Patients without progression at first response evaluation will continue treatment for a maximum of 9 months.

SUMMARY:
The aim of this study is to define a dose recommendation of vorinostat in pediatric oncology, to determine pharmacokinetics of vorinostat in children, determine response rates, safety and feasibility.

DETAILED DESCRIPTION:
Relapsed or progressive solid tumors and leukemias have a very poor prognosis in children despite intense multimodal treatment protocols involving polychemotherapy, surgery, and radiation. Therefore, innovative treatment strategies targeting specific molecular mechanisms are urgently required. A novel class of compounds with promising anti-tumoral activities is histone deacetylase (HDAC)-inhibitors. HDACs are key enzymes involved in regulation of chromatin-structure and function of several proteins, and aberrant activities of HDACs are found in many cancer cells. Pharmacological inhibition of HDACs causes cell cycle arrest, apoptosis, differentiation, inhibition of clonogenic growth, and anti-angiogenic effects in numerous cancer cells. In addition, promising anti-tumoral activity has been shown in several pre-clinical pediatric tumor models such as neuroblastoma, medulloblastoma, glioblastoma, retinoblastoma, rhabdomyosarcoma, osteosarcoma, Ewing's sarcoma, ATRT, and acute lymphoblastic leukemia. Several HDAC inhibitors are now in Phase I-III clinical trials in adult patients demonstrating a good safety profile and promising anti-neoplastic activity. The first of these compounds, suberoylanilide hydroxamic acid (SAHA, vorinostat, Zolinza), was recently approved by the FDA for the treatment of refractory cutaneous T-cell lymphoma. Vorinostat showed linear pharmacokinetics, good oral bioavailability and a broad range of anti-tumor activity in a Phase I clinical trial including 73 adult relapsed tumor patients. The determined peak plasma levels were in the range of 658±439 ng/ml (corresponding to 2.5±1.7 µM). At these concentrations, anti-tumoral effects on pediatric cancer cells and leukemias have been documented in vitro. Furthermore, vorinostat passes the blood brain barrier in mice, thus making it a suitable compound for the treatment of brain tumors.

The aim of this study is to define a dose recommendation of vorinostat in pediatric oncology, to determine pharmacokinetics of vorinostat in children, determine response rates, safety and feasibility. The design is an open, multicenter Phase I/II trial. Children and adolescents (3-18 years) with relapsed or therapy-refractory solid tumor, lymphoma or leukemia following standard treatment protocols in pediatric oncology will be included. 50 patients will be recruited over 2 years. Vorinostat will be taken orally once per day on an outpatient basis and the dose will be escalated until the individual maximum tolerated dose is established. This dose will then be applied for 3 months, when tumor response will be evaluated. Patients without progression at first response evaluation will continue treatment for a maximum of 9 months. After end of treatment (EOT) follow-up evaluations will be performed for 3 months. Pharmacokinetic studies will be performed in plasma, and in optional cerebrospinal fluid samples. Biomarkers (BMP4, IL-6, IL10 induction following Vorinostat treatment, basal histone acetylation, HDACs and H23B in archived tumor samples) will be determined and correlated with treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (3-18 years) with relapsed or therapy-refractory solid tumor, lymphoma or leukemia following standard first-line or relapse protocols in pediatric oncology
* Diagnosis confirmed by one of the Pathological, Radiological or Study Reference Centers recognized by the GPOH
* No other simultaneous anti-neoplastic treatment or radiation during the study and 1 months before enrolment
* Sufficient general condition (Lansky Score >50%)
* Life expectancy > 3 months
* Liver enzymes (ALT or AST) < 5x upper limit of normal reference value, bilirubin and creatinine < 3x upper limit of normal reference value
* Solid tumors: leukocytes > 2000/µl, thrombocytes > 50.000/µl and adequate bone marrow function to permit evaluations of hematopoietic toxicity
* No CTC grade 3 or 4 toxicity from previous treatments
* Normal ECG
* Written informed consent of the legal representatives and the patient if the patient is able to understand the study situation and to give consent (must be available before enrolment in the trial)
* Women with childbearing potential agree to use adequate contraception or to abstain from heterosexual activity throughout the study, starting with Visit 1.
* Sexually active male patient agrees to use an adequate method of contraception for the duration of the study
* Solid tumors: measurable disease activity according to RECIST criteria

Exclusion Criteria:

* History of deep vein thrombosis or pulmonary embolism
* Pregnancy and lactation
* Patient with concomitant treatments and/or anti-neoplastic treatment such as chemotherapy, immune therapy, and differentiation therapy, other targeted therapy, radiation. The use of valproic acid as prior antiepileptic therapy is allowed with a 30-day washout period.
* Prior exposure to Histone Deacetylase Inhibitors
* Known active HBV, HCV or HIV infection
* Patient with concomitant treatments such as amber [Hypericum perforatum], plant extracts, vitamins, and other anti-oxidative compounds
* Participation in other clinical trials or observation period of competing trials, respectively
* Patient is unable to swallow vorinostat suspension or capsules
* Patient on coumarin-derivative anticoagulants
* Any other medication which could accentuate known dose-dependent adverse effects of the study drug, for instance bone marrow depression or QT-prolongation

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
To determine a safe dose recommended (SDR) for the routine application of oral vorinostat (involving dose escalation) in children and adolescents (3-18 years) with relapsed/refractory solid tumor, lymphoma or leukemia. | After finding the individual MTD this dose will be applied for 3 months. Patients without progression at first response evaluation will continue treatment for a maximum of 9 months.
  A SDR is defined as the highest dose with no ≥ grade 3 toxicity according to CTC criteria (Dose Limiting Toxicity) in no more than 1/50 patient in this study.
  Dose Limiting Toxicity (DLT) is defined as any grade 3 or 4 toxicity according the CTCAE version 4.0 and judged by the investigator as definitely, probably or possibly related to the study drug.
  However, all DLTs will be subject to a second assessment by the Coordinating Investigator or a designated person.

SECONDARY OUTCOMES:
pharmacokinetics | d 8, when maximum tolerated dose (MTD) ist reached and after 3 months treatment at MTD
  Quantification of vorinostat concentration by mass spectrometry and enzymatically (AUC, Cmax, Cmin, tmax, Clearance, and t1/2).
  The pharmacokinetic study will investigate the correlation between dose administered, plasma concentration, CSF concentrations, intracellular inhibition of HDAC activity and glucuronosyltransferase polymorphisms as well as observed treatment responses and toxicities.
  Additionally:Intracellular HDAC activity in leukocytes using a fluorescence based enzymatic assay
antitumor effectiveness | three months after start of treatment with the individual MTD
  antitumor effectiveness of vorinostat as measured by treatment response rate
association of the histone deacetylase (HDAC)-inhibiting activity with the dose administered, toxicity, and treatment response | d8, after reaching the MTD and after 3 months treatment at MTD
  Intracellular vorinostat concentrations and pharmacologic target (HDAC) inhibition in peripheral leukocytes will be determined as a pharmacodynamic surrogate parameter. The latter assay is based on conversion of a fluorigenic acetyl-substrate by the enzymatic activity of HDACs which is specifically inhibited by vorinostat in a concentration dependent manner. The performance of the assay in patient plasma samples has been validated according to the FDA recommendations "Guidance for Industry Bioanalytical Method Validation".
safety | during dose escalation and during 3 months treatment at MTD every week; during prolongation of treatment and follow-up every second week
  The analysis of safety assessments will include summaries of the following categories of safety and tolerability data collected for each subject:
  * Drug Exposure(s)
  * Adverse Events (AEs and SAEs, AEs leading to withdrawal)
  * Clinical Laboratory Investigations
  * Hemodynamics (vital signs)
  * ECG Investigations
  Frequencies of patients experiencing at least one AE will be displayed. Severity of the AEs will be graded according to the CTCAEv4.0. Summary tables will present the number of patients observed with AEs, the corresponding percentages and 95% CI.
duration of response in responding patients | every 3 months until progression of tumor
  MRI and MIBG (in case of neuroblastoma)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Witt, Prof. Dr., Principal Investigator — University Hospital Heidelberg and German Cancer Research Center (DKFZ)
Locations (10):
- Germany (10):
  - Clinic for Pediatric Oncology, Hematology, Immunology and Clinical Cooperation Unit Pediatric Oncology, Heidelberg, Baden-Wurttemberg
  - Childrens's Hospital, Pediatric Oncology and Hematology, Augsburg
  - Prof. Hess Childrens's Hospital, Pediatric Oncology and Hematology, Bremen
  - University Children's Hospital, Pediatric Oncology and Hematology, Cologne
  - University Childrens's Hospital, Pediatric Oncology and Hematology, Essen
  - University Children's Hospital, Clinic IV, Freiburg im Breisgau
  - Department of Pediatric Oncology and Hematology University Hospital Eppendorf (UKE), Hamburg
  - University Children's Hospital, Pediatric Oncology and Hematology, MHH, Hanover
  - University Childrens's Hospital, Pediatric Oncology and Hematology, Jena
  - Department of Pediatric Oncology and Hematology University Children's Hospital, Münster

REFERENCES:
- [Derived] van Tilburg CM, Milde T, Witt R, Ecker J, Hielscher T, Seitz A, Schenk JP, Buhl JL, Riehl D, Fruhwald MC, Pekrun A, Rossig C, Wieland R, Flotho C, Kordes U, Gruhn B, Simon T, Linderkamp C, Sahm F, Taylor L, Freitag A, Burhenne J, Foerster KI, Meid AD, Pfister SM, Karapanagiotou-Schenkel I, Witt O. Phase I/II intra-patient dose escalation study of vorinostat in children with relapsed solid tumor, lymphoma, or leukemia. Clin Epigenetics. 2019 Dec 10;11(1):188. doi: 10.1186/s13148-019-0775-1. PMID 31823832
- [Derived] Witt O, Milde T, Deubzer HE, Oehme I, Witt R, Kulozik A, Eisenmenger A, Abel U, Karapanagiotou-Schenkel I. Phase I/II intra-patient dose escalation study of vorinostat in children with relapsed solid tumor, lymphoma or leukemia. Klin Padiatr. 2012 Oct;224(6):398-403. doi: 10.1055/s-0032-1323692. Epub 2012 Aug 22. PMID 22915450